CLINICAL TRIAL: NCT00576264
Title: Peritoneal Cavity Derived Stem Cells: A Pilot Study
Brief Title: Stem Cells Found in the Abdominal Cavity in Humans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Prediman Krishnan Shah, MD, Cedars-Sinai Medical Center
Other Study IDs: 11388
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-12

CONDITIONS: Intra-abdominal Surgery
Keywords: open abdominal surgery; abdominal laparoscopic surgery; peritoneal stem cells; patients scheduled for any type of elective intra-abdominal surgery at Cedars-Sinai Medical Center with designated surgeons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peritoneal fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to determine the genotype (genetic composition) and phenotype (physical appearance) of cells derived from the abdominal cavity to determine whether stem cells are present.

DETAILED DESCRIPTION:
The purpose of this study is to determine the presence and characterization of stem cells in human peritoneal cavity. Peritoneal lavage fluid from patients who undergo elective open abdomen will be collected for this purpose. Peritoneal lavage is normally a routine part of abdominal surgical procedure and usually is discarded after surgery. The patient will undergo surgical procedure as usual and there will be no added procedures during surgery.

This study will collect and analyze peritoneal fluid for the existence and characteristics of stem cells from 15 patients undergoing scheduled elective intra-abdominal surgery by designated surgeons at Cedars-Sinai Medical Center. The types of abdominal surgery could be open abdominal surgery or laparoscopic surgery. Peritoneal washing is routinely done in abdominal surgeries. We will collect these fluids to analyze whether stem cells exist in human peritoneal cavity. The fluids will be collected in a sterile fashion. The collected fluid will be further processed in the laboratory for the purpose of the study.

Medical record review will be conducted. Information collected will include age, gender, past and current medical history, current indication for intra-abdominal surgery, substance exposure history, medication history which will be obtained from review of patients' medical records. The information will be maintained using coded entry and there will be no link between patient identifiers to the study codes.

ELIGIBILITY:
Inclusion Criteria:

1. 20-60 years old
2. Male or females who are scheduled to undergo elective abdomen surgery

Exclusion Criteria:

1. Minors
2. Pregnant women
3. Known personal or family history of genetic disorders
4. Known history of malignancy
5. Known history of advanced liver or renal disease
6. HIV Positive: only patients who have tested negative during routine testing of their donated blood prior to surgery will be included in the study.
7. Hepatitis B and C positive
8. Scheduled to undergo lap banding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: subjects undergoing scheduled elective intra-abdominal surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-04; Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Prediman K Shah, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States